CLINICAL TRIAL: NCT06312332
Title: Michigan Emergency Department Improvement Collaborative (MEDIC) AltERnaTives to Admission for Pulmonary Embolism
Brief Title: Michigan Emergency Department Improvement Collaborative (MEDIC) Alert; Pulmonary Embolism (PE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Geoffrey Barnes, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00220089; 1R01HL163438-01A1 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism
Keywords: Emergency Department
MeSH Terms: conditions — Pulmonary Embolism; Emergencies | interventions — Emergency Service, Hospital

STUDY DESIGN:
Intervention Model Description: cluster-randomized stepped-wedge design with two or more sites assigned at each of four steps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEDIC site (Experimental)
  Interventions: Behavioral: Pulmonary Embolism (PE) Care in Emergency Department (ED)

INTERVENTIONS:
Behavioral: Pulmonary Embolism (PE) Care in Emergency Department (ED) — Utilize implementation mapping to facilitate intervention development and evaluation that can be disseminated broadly in diverse settings. Intervention to include a structured education program for clinicians on home management of patients with low-risk PE led by regional/national leaders, the development of Clinician pre-commitment, point-of-care nudge including a clinical guideline integrated into an electronic health record clinical decision support, facilitated medication access, and dedicated outpatient rapid-follow up.

SUMMARY:
This study is a quality improvement project to evaluate health care management of pulmonary embolism (PE) patients. The researchers are testing an intervention to determine if it prevents unnecessary hospital admissions.

DETAILED DESCRIPTION:
The study team anticipates that there will be 5800 acute PE patients over multiple sites.

ELIGIBILITY:
Inclusion Criteria:

* Participation in MEDIC collaborative
* Identified site physician champion
* Annual volume of acute PE ≥80 (measured in 2022)

Exclusion Criteria:

* Pediatric-only hospital/ED
* No site physician champion identified
* Annual volume of acute PE <80 (measured in 2022)
* Existing formal clinical pathway for outpatient management of low-risk PE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of patients discharged home from Emergency Department (ED) | 3 months Pre-intervention, Up to 18 months Post-intervention
  Reported by participating center indicating the proportion of patients discharged home from ED

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Barnes, Study Chair — University of Michigan
Locations (1):
- Michigan Emergency Department Improvement Collaborative partners, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith SN, Greineder CF, Errickson J, Burns J, Seagull FJ, Kocher KE, Kline JA, Kullgren JT, Lanham MSM, Krein SL, Barnes GD. A stepped wedge cluster randomized implementation trial to increase outpatient management of low-risk pulmonary embolism from the emergency department - the MEDIC ALERT PE study. Implement Sci Commun. 2025 Apr 2;6(1):33. doi: 10.1186/s43058-025-00720-1. PMID 40176133